CLINICAL TRIAL: NCT05732818
Title: Clinical Investigation Plan First in Human Trial Lumbar Operatively Inserted PerQdisc Artificial Implant Following Nuclectomy "LOPAIN3"
Brief Title: Lumbar Operatively Inserted PerQdisc Artificial Implant Following Nuclectomy 3
Acronym: LOPAIN3
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended as enrollment of patients was difficult and no participants could be found for two years.
Sponsor: Spinal Stabilization Technologies (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPQ114.B: LOPAIN3
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Back Pain With Radiation; Radiculopathy; Back Pain; Disc Herniation; Herniated Nucleus Pulposus; Herniated Disc; Disc Injury; Disk Herniated Lumbar
MeSH Terms: conditions — Back Pain; Radiculopathy; Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Patients will receive one implant if they meet all inclusion/exclusion criteria after a review by the Medical Advisory Board (MAB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar Disc Nucleus Replacement following discectomy (Experimental): All patients meeting all inclusion criteria and no exclusion criteria will be considered for nucleus replacement surgery following a review by the Medical Advisory Board.
  Interventions: Device: PerQdisc Nucleus Replacement System

INTERVENTIONS:
Device: PerQdisc Nucleus Replacement System — Lumbar spine disc nucleus replacement system. All patients meeting all inclusion criteria and no exclusion criteria will be considered for nucleus replacement surgery following a review by the Medical Advisory Board.

SUMMARY:
This study is a First in Human, prospective, multi-center clinical study intended to collect safety and performance information for the Spinal Stabilization Technologies PerQdisc® Nucleus Replacement System and procedure concurrently following a successful discectomy using a minimally invasive posterolateral (MIPL) approach. Patients that are at least 21 years or older, presenting with symptomatic radiculopathy from a focal lumbar disc herniation that requires surgical decompression will be included in this study.

DETAILED DESCRIPTION:
The PerQdisc® Nucleus Replacement System is comprised of an in situ formed silicone-based prosthesis with its delivery system, implant fill device, dispenser gun, a disc access system and two different imaging balloons. For this trial, the PerQdisc® will be implanted using minimally invasive posterolateral (MIPL) approach. The implanted device provides an effective means of replacing dysfunctional nucleus pulposus while supporting the native annulus fibrosis to bridge annular defects.

Patients that suffer clinically significant lumbar disc herniations currently undergo discectomy procedures to relieve nerve root compression. The standard discectomy procedure does not correct the annular defect associated with the herniation and is associated with a risk for re-herniation. In addition, the progressive loss of disc height and overall lack of disc turgor and weight bearing capacity is thought to be associated with downstream degenerative changes that may lead to chronic low back pain and premature spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature and at least 21 years of age.
* Patient has a lumbar disc herniation, between L1-S1, with compressive radiculopathy of the traversing nerve root requiring partial discectomy or sequestrectomy. Only one lumbar disc may be treated with the PerQdisc device.
* Patient must have an overall disc herniation (extrusion or protrusion) such that half or less of the width of the dorsal annulus of the spinal canal, is affected by the herniation. The width of the canal is defined by the lateral recesses and the central canal (i.e. pedicle to pedicle).
* Patient must have a minimum of 6 mm of disc height as measured in the center of the affected disc.
* Patient is willing and able to give informed consent.
* All surgeries must be approved by at least 2 members of the Medical Advisory Board (MAB) - potential anatomical limitations of safely accessing Kambin's, extent of annular disruption, as well as overall patient criteria will be evaluated

Exclusion Criteria:

* Patient has had prior lumbar spine surgery at the index level (nucleoplasy is acceptable).
* Patient has had spinal fusion in the lumbar spine. Cervical or thoracic fusion is allowed as long as there are no neurologic deficits in the lower extremities.
* Patient has spondyloarthropathy or other spondylolisthesis greater than 4 mm or spondylolysis at the index level (on standing X-ray).
* Patient has underlying moderate or severe spinal stenosis (congenital, degenerative, or due to epidural lipomatosis) at any level. If the index level shows stenosis due to the disc herniation, it is acceptable if the index level is going to be treated concurrently with the PerQdsic procedure.
* Patient has compressive radiculopathy of the exiting nerve root at the index level.
* Patient has significant facet disease. Significant is defined as clinically confirmed by diagnostic block or radiologically grade 2 or higher (mild joint narrowing and irregularity are acceptable, but not sclerosis or osteophyte formation).
* Patient has any known active malignancy.
* Patient has previously undergone or currently on immunosuppressive therapy. Steroids used to treat inflammation are allowed.
* Patient has active local or systemic infection.
* Patient has been diagnosed with hepatitis, rheumatoid arthritis, lupus erythematosus, or other autoimmune disease including AIDS, AIDS related complex (ARC) and HIV.
* Patient has diabetes mellitus (Type 1 or 2) requiring daily insulin management.
* Patient has osteopenia of the spine (T-score of -1.0 or lower). All patients 50 years of age or older, and any post menopausal women with a history of fractures should have a dual x-ray absorptiometry (DEXA) scan to confirm exclusion.
* Patient has morbid obesity defined as a body mass index (BMI) more than 35 (>35).
* Patient has a known allergy to silicone or barium sulfate.
* Patient has a broad disc herniation that is wider than ½ of the dorsal annulus forming the wall of the spinal canal
* Patient requires decompression involving disruption of the midline bony-ligamentous elements (i.e. laminectomy).
* Patient has a significant Schmorl's node at the level to be treated, or any Schmorl's nodes affecting 3 or more lumbar levels. Significant is defined as a large, rectangular or irregular shaped node that has an associated active inflammatory process (Modic I changes).
* Patient has more than 20 degrees of mobility on flexion/extension radiographs at the index level
* Patient has more than 10 degrees of lumbar scoliosis.
* Patient belongs to a vulnerable population or has a condition such that his/her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g. developmentally disabled, prisoner, chronic alcohol/ substance abuser)
* Patient is pregnant or plans to become pregnant during the course of the study. Pregnancy ruled out by serum HCG. If patient becomes pregnant during the course of the study and wishes to continue study participation, a new Pregnancy Informed Consent must be completed.

Intraoperative Exclusion:

* Poor radiological visualization of Kambin's triangle
* Patient has annular defect following surgical treatment of the disc herniation/protrusion that is greater than 6 mm
* Sustained irritation of the exiting nerve root during any aspect of the annular dilation technique (leg movement or if performing with electrical monitoring) in spite of repositioning instruments.
* Protrusion of the 50A Imaging Balloon up to or beyond the outer margin of the vertebra during the imaging steps.
* Patient has a violated endplate as determined by imaging balloons during fluoroscopy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Patients with Serious Adverse Events related to the PerQdisc | 12 months
  Freedom from device- and procedure-related serious adverse events definitely related to the PerQdisc Device or the PerQdisc Surgical Procedure

SECONDARY OUTCOMES:
Performance: ODI | 3 months
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient reported outcome tool
Performance: ODI | 6 months
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient reported outcome tool
Performance: ODI | 12 months
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient reported outcome tool
Performance: ODI | 24 months
  Change in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient reported outcome tool
Performance: VAS Back | 3 months
  Change in back pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Back | 6 months
  Change in back pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Back | 12 months
  Change in back pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Back | 24 months
  Change in back pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Leg | 3 months
  Change in leg pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Leg | 6 months
  Change in leg pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Leg | 12 months
  Change in leg pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: VAS Leg | 24 months
  Change in leg pain values as measured by the 100 millimeter Visual Analog Scale (VAS)
Performance: Analgesic Score | 3 months
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale from 0 (no meds) to 4 (high dose opioids)
Performance: Analgesic Score | 6 months
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale from 0 (no meds) to 4 (high dose opioids)
Performance: Analgesic Score | 12 months
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale from 0 (no meds) to 4 (high dose opioids)
Performance: Analgesic Score | 24 months
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale from 0 (no meds) to 4 (high dose opioids)
Safety: Number of Patients with Reherniation/recurrent disc herniation | 3 months
  Freedom from reherniation/recurrent disc herniation
Safety: Number of Patients with Reherniation/recurrent disc herniation | 6 months
  Freedom from reherniation/recurrent disc herniation
Safety: Number of Patients with Reherniation/recurrent disc herniation | 12 months
  Freedom from reherniation/recurrent disc herniation
Safety: Number of Patients with Reherniation/recurrent disc herniation | 24 months
  Freedom from reherniation/recurrent disc herniation
Safety: Number of Patient that Received Supplemental fixation | 3 months
  Freedom from supplemental fixation at the index level(s) including basivertebral nerve ablation, radiofrequency ablation or spinal cord stimulator
Safety: Number of Patient that Received Supplemental fixation | 6 months
  Freedom from supplemental fixation at the index level(s) including basivertebral nerve ablation, radiofrequency ablation or spinal cord stimulator
Safety: Number of Patient that Received Supplemental fixation | 12 months
  Freedom from supplemental fixation at the index level(s) including basivertebral nerve ablation, radiofrequency ablation or spinal cord stimulator
Safety: Number of Patient that Received Supplemental fixation | 24 months
  Freedom from supplemental fixation at the index level(s) including basivertebral nerve ablation, radiofrequency ablation or spinal cord stimulator

OTHER OUTCOMES:
Exploratory Endpoint: Disch Height | 3 months
  Disc height in millimeters at each clinical visit as measured on plain film X-ray
Exploratory Endpoint: Disch Height | 6 months
  Disc height in millimeters at each clinical visit as measured on plain film X-ray
Exploratory Endpoint: Disch Height | 12 months
  Disc height in millimeters at each clinical visit as measured on plain film X-ray
Exploratory Endpoint: Disch Height | 24 months
  Disc height in millimeters at each clinical visit as measured on plain film X-ray
Exploratory Endpoint: RoM | 3 months
  Preservation of range of movement (expressed in degrees) at the index and adjacent levels at baseline compared to follow-up using flexion/extension radiographs
Exploratory Endpoint: RoM | 6 months
  Preservation of range of movement (expressed in degrees) at the index and adjacent levels at baseline compared to follow-up using flexion/extension radiographs
Exploratory Endpoint: RoM | 12 months
  Preservation of range of movement (expressed in degrees) at the index and adjacent levels at baseline compared to follow-up using flexion/extension radiographs
Exploratory Endpoint: RoM | 24 months
  Preservation of range of movement (expressed in degrees) at the index and adjacent levels at baseline compared to follow-up using flexion/extension radiographs
Exploratory Endpoint: Neurological Status | 3 months
  Maintenance and/or improvement of baseline neurologic status through physical assessment evaluating nerve compression at baseline and post-surgical follow-up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale
Exploratory Endpoint: Neurological Status | 6 months
  Maintenance and/or improvement of baseline neurologic status through physical assessment evaluating nerve compression at baseline and post-surgical follow-up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale
Exploratory Endpoint: Neurological Status | 12 months
  Maintenance and/or improvement of baseline neurologic status through physical assessment evaluating nerve compression at baseline and post-surgical follow-up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale
Exploratory Endpoint: Neurological Status | 24 months
  Maintenance and/or improvement of baseline neurologic status through physical assessment evaluating nerve compression at baseline and post-surgical follow-up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale

CONTACTS AND LOCATIONS:
Locations (2):
- Sanatorio Americano, Asunción, Paraguay
- Republican Specialized Scientific Practical Medical Center of Endocrinology named after Academician Y.Kh. Turakulova, Tashkent, Tashkent, Uzbekistan